CLINICAL TRIAL: NCT00342498
Title: Estrogen Receptor Gene Mutations
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999994012; OH94-E-N012
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-17

CONDITIONS: Mutations; Hormones
Keywords: DNA; Hormone; Resistance; Skeleton

SUMMARY:
We propose to analyze a DNA sample for mutations in the estrogen receptor gene from a patient who appears insensitive to estrogen hormone treatment.

DETAILED DESCRIPTION:
We propose to analyze a DNA sample for mutations in the estrogen receptor gene from a patient who appears insensitive to estrogen hormone treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patient is individual with estrogen insensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1994-01-12; Study Completion 2008-06-17

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio